CLINICAL TRIAL: NCT04263675
Title: Human Milk: Understanding the Mechanisms Linked to the Prevention of Obesity and Diabetes in Children Exposed in Utero to Gestational Diabetes
Acronym: LAIT-M
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Julie Robitaille, Principal investigator, Laval University
Other Study IDs: LAIT-M
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM+: Women with history of gestational diabetes
- GDM-: Women without history of gestational diabetes

SUMMARY:
Breastfeeding has been associated with decreased obesity. However, this relationship is not as clear in children who have been exposed to GDM and the mechanisms involved are little known. The overall objective of the project is to study the mechanisms of breastfeeding on the growth of children in women who have had a GDM. More specifically, the project want to compare the macronutrient and hormone composition of breast milk of women with and without GDM. Investigators also want to associate the levels of hormones related to satiety and energy metabolism (i.e. endocannabinoids, ghrelin, leptin) in the human milk of women with or without DG and the growth of the child. A total of 60 women (30 with GDM and 30 without GDM) will collect breastmilk at 2 months postpartum.

DETAILED DESCRIPTION:
Other data collected:

Waist circumference, DXA, Fasted blood sample, Oral glucose tolerance test, Breastfeeding habits, Food habits, Baby's height et weight.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding women

Exclusion Criteria:

* Type 1 or type 2 diabetes
* Preterm birth
* History of bariatric surgery
* Multiple births

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with or without GDM
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Study the mechanisms linked to the effect of breastfeeding on the growth of children in women who have had GDM. | 2 years

SECONDARY OUTCOMES:
Compare macronutrient and hormone composition of breast milk of women with and without GDM. | 6 months
Associate level of hormones related to satiety and energy metabolism (i.e. endocannabinoids, ghrelin, leptin) in the human milk of women with or without GDM and the growth of the child. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petitclerc I, Perron J, Dugas C, Mayer T, Raymond F, Di Marzo V, Veilleux A, Robitaille J. Association between gestational diabetes mellitus, maternal health and diet, and gut microbiota in mother-infant dyads. BMC Pregnancy Childbirth. 2025 Apr 24;25(1):486. doi: 10.1186/s12884-025-07584-2. PMID 40275186
- [Derived] Fradet A, Castonguay-Paradis S, Dugas C, Perron J, St-Arnaud G, Marc I, Doyen A, Flamand N, Dahhani F, Di Marzo V, Veilleux A, Robitaille J. The human milk endocannabinoidome and neonatal growth in gestational diabetes. Front Endocrinol (Lausanne). 2024 Jun 13;15:1415630. doi: 10.3389/fendo.2024.1415630. eCollection 2024. PMID 38938519